CLINICAL TRIAL: NCT00404963
Title: A Single-Blind, Randomized, Placebo Controlled, Ascending Single and Repeat Dose Study With Once Daily Dosing to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GSK376501 and to Evaluate Food Effects and the Relative Bioavailability of a Tablet Formulation Compared to the Powder for Reconstitution Formulation in Healthy Overweight and Obese Subjects (DIX109177)
Brief Title: A Study To Investigate The Safety And Metabolism Of GSK376501 In Overweight Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DIX109177
Record Dates: First submitted 2006-11-27; First posted 2006-11-29 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: GSK376501,; First Time in Human,; Single Dose,; Dose Escalation,; Healthy Overweight/Obese Volunteer
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: placebo
Drug: GSK376501
  Other Names: placebo

SUMMARY:
This study represents the first administration of GSK376501 in humans and the goal is to evaluate its initial safety and tolerability. The way the human body processes GSK376501 will also be determined.

DETAILED DESCRIPTION:
A Single-Blind, Randomized, Placebo Controlled, Ascending Single and Repeat Dose Study with Once Daily Dosing to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GSK376501 and to Evaluate Food Effects and the Relative Bioavailability of a Tablet Formulation Compared to the Powder for Reconstitution Formulation in Healthy Overweight and Obese Subjects (DIX109177)

ELIGIBILITY:
Inclusion:

* Healthy
* Non-smoking
* Overweight or obese subjects with a BMI between 27 and 35.

Exclusion:

* Women who are pregnant, lactating, or are of child-bearing potential

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-10; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Safety will be monitored by assessing adverse reactions,changes in laboratory values (hematology, clinical chemistry, urinalysis),changes in vital signs (oral body temperature,60 second respiratory rate, blood pressure and heart rate), and ECG changes. | throughout the study

SECONDARY OUTCOMES:
Blood levels of GSK376501 Effects of GSK376501 on the body, by measuring changes in insulin, glucose, and other markers | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, MPH, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Evansville, Indiana, United States